CLINICAL TRIAL: NCT05398432
Title: The Effect of Self-Care Supported Motivational Interviewing on Patients' Self-Care Strength and Disease Adjustment in Patients Receiving Hemodialysis Treatment
Brief Title: The Effect of Hemodialysis Treatment on Self-Care Power and Disease Adjustment of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdullah Gerçek (Other)
Responsible Party: Sponsor-Investigator, Abdullah Gerçek, lecturer, Muş Alparslan University
Organization: Muş Alparslan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUŞ ALPARSLAN UNIVERSITY
Record Dates: First submitted 2021-09-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Motivation; Hemodialysis Complication; Patient Compliance
Keywords: hemodialysis; self care; motivational interview
MeSH Terms: conditions — Patient Compliance | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: randomized controlled trial design
Masking Description: Randomization was performed to ensure that any observed changes in outcomes between the experimental and control groups were free from bias. Four sessions in the hemodialysis unit were listed and four lots were drawn by a person who was unaware of the study. The first draw was the experimental group, the second draw was the control group, the third draw was the experimental group, and the fourth draw was the control group. Thus, the patients in the morning and afternoon sessions on Monday-Wednesday-Friday constituted the control group, and the patients in the Tuesday-Thursday-Saturday morning and afternoon sessions constituted the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Experimental): The control group did not intervene
  Interventions: Other: motivational interview
- experiment (Experimental): Initial data were collected after meeting the patients. Then, a total of 6 seans, 1 seans per week, were performed on the patients. Self-care training was given in the 1st, 2nd and 3rd seans. Motivational interviews were conducted in the 4th, 5th and 6th seans. After the first seans of the self-care supported motivational interview, the "Self Care and Adaptation Training Guide" prepared by the researcher in line with the literature was given to the experimental group. Second data were collected from patients after 6 weeks. Follow-up data were collected for 4 weeks without any intervention.
  Interventions: Other: motivational interview

INTERVENTIONS:
Other: motivational interview — After the pre-test data were applied to all patients, before starting the motivational interview seans, the patients were informed about the interview intervals, duration, and how many times they would be held. In the second week, motivational interview seans were started with the patients. seans with patients took place during the hemodialysis seans. A total of 6 seans were held, one seans per week. After the first seans of the self-care supported motivational interview, the "Self-Care and Adaptation to Disease Training Guide" prepared by the researcher in line with the literature was given to the experimental group. Self-care training was given in the first, second and third seans. Motivational interviews were conducted in the fourth, fifth and sixth seans. Motivational interviewing techniques were used for patients to realize their self-care activities. seans were held individually with the patients and each seans lasted approximately 15-20 minutes.

SUMMARY:
The study was conducted to determine the effect of self-care supported motivational interviewing on patients receiving hemodialysis treatment on self-care power, disease compliance and metabolic variables.

The study was completed with 77 patients. In the collection of data; Personal Information Form, Self-Care Strength Scale, Chronic Disease Adjustment Scale and Patient-Specific Metabolic Variables Form were used.

DETAILED DESCRIPTION:
The study was conducted as a randomized controlled, repeated measurement, experimental research design.

The research was carried out in Muş Provincial Health Directorate Muş State Hospital Hemodialysis Unit between October 2020 and March 2021. There are 6 nurses, 7 dialysis technicians, 5 assistant health personnel, 2 specialist physicians, 28 patient beds and 28 hemodialysis machines in the hemodialysis unit where the research was conducted. In the hemodialysis unit, there are 1 waiting room where patients and their attendants wait, 4 private rooms and 2 large halls where patients receive hemodialysis treatment. There is no attempt at motivational interviewing in the hemodialysis center where the research was conducted.

The population of the study consisted of 97 patients who received hemodialysis treatment at the Muş Provincial Health Directorate, Muş State Hospital, Hemodialysis Unit on the specified dates. The sample of the research is "G. Using the "Power-3.1.9.2" program and based on similar articles, 80% power was determined at an effect size of 0.70 and it was calculated to have a minimum of 68 subjects in total. In the hemodialysis unit where the research was conducted, 85 patients who met the research criteria and volunteered to participate in the research were formed because 2 patients did not attend hemodialysis treatment regularly, 4 patients did not want to participate in the study, 3 patients had poor general health conditions, 2 patients had hearing problems, and 1 patient was transferred to another dialysis center. . Using the simple random sampling method, 45 patients were assigned to the experimental group and 40 patients to the control group. However, during the research period, the study was completed with 37 patients in the control group, as 40 patients in the experimental group and 3 patients in the control group died due to the death of 2 patients from the experimental group, the death of 2 patients and the transfer of 1 patient to another hemodialysis center during the research period.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving hemodialysis treatment for at least three months at the time of the study,
2. HD treatment for 3-4 hours 2 or 3 days a week,
3. 18 years old and above,
4. Open to communication and cooperation,
5. Not visually or hearing impaired,
6. Being a reader and writer,
7. Not having any psychiatric diagnosis and/or not using any psychiatric medication,
8. Have not received motivational interviewing training before,
9. Individuals who agreed to participate in the study were included in the study.

Exclusion Criteria:

1. who are under the age of 18,
2. Having a communication problem,
3. Individuals who did not want to participate in the study or did not want to continue were excluded from the study.ı

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
self care power scale | 6 week
  ıt is a scale used to measure an invidual's self-care abilit. the maximum score is 140. the hiğher the score obtained from the scale indicates the hiğh level of self-care ability and power of the invidual.

SECONDARY OUTCOMES:
Chronic Disease Adjustment Scale | 6 week
  The scale was developed to measure the level of compliance of individuals with chronic diseases. The total score that can be obtained from the scale is 125. An increase in the scores obtained from the sub-dimensions and/or the whole scale means that the patients' level of compliance with the disease also increases.

CONTACTS AND LOCATIONS:
Overall Officials: abdullah gerçek, doktora, Principal Investigator — Muş Alparslan University; serap parlar kılıç, Study Director — Inonu University
Locations (1):
- Mus State Hospital, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no, not shared with other people